CLINICAL TRIAL: NCT00535938
Title: MDs on Botox Utility (MOBILITY)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: AGN/MMC B00705
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Blepharospasm; Torticollis; Strabismus; Muscle Spasticity
MeSH Terms: conditions — Blepharospasm; Torticollis; Strabismus; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Naïve to Botox® treatment: Initiating treatment with BOTOX® upon entry to the project.
  Interventions: Other: botulinum toxin type A
- Non-naïve to Botox® treatment: Receiving ongoing treatment with BOTOX® upon entry to the project.
  Interventions: Other: botulinum toxin type A

INTERVENTIONS:
Other: botulinum toxin type A — There will be no protocol-mandated intervention with regard to physician treatment choice or management of patient condition once the patient is enrolled in the project.

SUMMARY:
The MOBILITY Project is a prospective, non-randomized, observational, multi-centre evaluation of Health Utility via the SF-12® Health Survey Scores and the SF-6D in patients receiving BOTOX® for therapeutic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for BOTOX® treatment deemed medically necessary by their physician
* Patient (and/or patient's authorized legal representative) should provide written informed consent; a patient under the age of 18 must review and sign the Patient Assent Form
* Patients at the age of or over 14

Exclusion Criteria:

* Patient is participating in a clinical trial for any BOTOX® indication
* Patient with any contraindications to use botulinum toxin A

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 1372 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Started | 506 | 866
Completed | 115 | 404
Not Completed | 391 | 462

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment | Total
Number analyzed (Participants) | 506 | 866 | 1372
Age, Customized [Number; unit: Participants]
  14 to 17 years | 22 | 28 | 50
  18 to 65 years | 374 | 641 | 1015
  >65 years | 110 | 197 | 307
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 577 | 881
  Male | 202 | 289 | 491

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Cervical Dystonia
Description: Cervical dystonia is a condition in which the neck muscles contract involuntarily, causing the head to turn to one side, forward or backward. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 505 days for patients with cervical dystonia.
Time Frame: Baseline, SV1 (up to 505 days)
Population: Efficacy Cohort: all enrolled patients who had a valid SF-6D score at baseline and at least one valid SF-6D score at a subsequent visit within the prospective period and who had data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 44 | 186
Scores on a Scale
  Baseline | 0.650 (0.154) | 0.676 (0.143)
  Change from Baseline at SV1 (N=33,174) | 0.020 (0.084) | -0.001 (0.104)

2. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Blepharospasm
Description: Blepharospasm is a condition in which the eyelids blink/close involuntarily. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 542 days for patients with blepharospasm.
Time Frame: Baseline, SV1 (up to 542 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 23 | 56
Scores on a Scale
  Baseline | 0.718 (0.122) | 0.754 (0.132)
  Change from Baseline at SV1 (N=21, 51) | 0.053 (0.156) | 0.014 (0.120)

3. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Hyperhidrosis
Description: Hyperhidrosis is a condition causing excessive sweating, regardless of temperature or exercise. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 1,273 days for patients with hyperhidrosis.
Time Frame: Baseline, SV1 (up to 1,273 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 101 | 107
Scores on a Scale
  Baseline | 0.782 (0.129) | 0.799 (0.115)
  Change from Baseline at SV1 (N=58, 60) | 0.010 (0.136) | -0.000 (0.124)

4. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Cerebral Palsy
Description: Cerebral Palsy is a disability resulting in muscular incoordination and speech disturbances. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 925 days for patients with cerebral palsy.
Time Frame: Baseline, SV1 (up to 925 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 3 | 15
Scores on a Scale
  Baseline | 0.712 (0.131) | 0.733 (0.117)
  Change from Baseline at SV1 (N=0, 8) | NA (NA) — No patients had data at this time point. | 0.018 (0.114)

5. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Adult Focal Spasticity
Description: Adult Focal Spasticity is a condition in which muscles are continuously tight or stiff in a certain area. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 1,562 days for patients with adult focal spasticity.
Time Frame: Baseline, SV1 (up to 1,562 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 149 | 241
Scores on a Scale
  Baseline | 0.621 (0.111) | 0.635 (0.124)
  Change from Baseline at Week 4 (N=114, 201) | 0.002 (0.096) | 0.008 (0.096)

6. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With Facial Nerve Disorder
Description: Facial nerve disorder is a condition causing twitching, weakness or paralysis of the face. The SF-12 consists of 12 questions on various health questions. Health utility is a numerical indicator of a person's preferences for a given health state or health outcome. Health utility is a sub-score ranging from 0 (death) to 1 (perfect health) and is calculated from the SF-12 total score based on the following items: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 765 days for patients with facial nerve disorder.
Time Frame: Baseline, SV1 (up to 765 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 38 | 77
Scores on a Scale
  Baseline | 0.770 (0.134) | 0.759 (0.134)
  Change from Baseline at SV1 (N=30, 63) | 0.035 (0.158) | 0.002 (0.111)

7. Primary Outcome: Change From Baseline in the SF-6D Measure Health Utility (Quality of Life) Score Using the SF-12® Questionnaire for Patients With "Other" Disorders
Description: "Other" disorders include focal dystonia (involuntary muscular contractions/abnormal postures), headache, pain, tics (sudden, repetitive, nonrhythmic movements/vocalizations), tremors (unintentional, rhythmic muscle movements), and other nonspecified disorders. The SF-12 is 12 questions on various health questions. Health utility is a numerical indicator of a person's preference for a given health state or health outcome. Health utility is a sub-score ranging from 0(death) to 1(perfect health) calculated from the SF-12 total score based on: physical functioning, role participation, social functioning, bodily pain, mental health, and vitality and is termed SF-6D. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The length of time between Baseline and SV1 is scheduled at the physician's discretion and was a maximum of 568 days for patients with "other" disorders.
Time Frame: Baseline, SV1 (up to 568 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 47 | 84
Scores on a Scale
  Baseline | 0.570 (0.137) | 0.610 (0.118)
  Change from Baseline at SV1 (N=33, 72) | 0.060 (0.086) | 0.028 (0.113)

8. Secondary Outcome: BOTOX® Dose in Patients With Cervical Dystonia
Description: Cervical dystonia is a condition in which the neck muscles contract involuntarily, causing the head to turn to one side, forward or backward. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 505 days for patients with cervical dystonia.
Time Frame: Baseline, SV1 (up to 505 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 48 | 202
Units
  Baseline | 154.8 (61.1) | 242.7 (99.6)
  SV1 (N=37, 187) | 169.9 (70.2) | 246.4 (101.7)

9. Secondary Outcome: BOTOX® Dose in Patients With Blepharospasm
Description: Blepharospasm is a condition in which the eyelids blink/close involuntarily. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 542 days for patients with blepharospasm.
Time Frame: Baseline, SV1 (up to 542 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 24 | 59
Units
  Baseline | 42.9 (13.8) | 67.3 (54.3)
  SV1 (N=23, 54) | 47.8 (22.7) | 61.9 (39.5)

10. Secondary Outcome: BOTOX® Dose in Patients With Hyperhidrosis
Description: Hyperhidrosis is a condition causing excessive sweating, regardless of temperature or exercise. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 1,273 days for patients with hyperhidrosis.
Time Frame: Baseline, SV1 (up to 1,273 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 151 | 137
Units
  Baseline | 192.5 (60.4) | 203.6 (74.8)
  SV1 (N=80, 97) | 186.9 (53.8) | 206.5 (81.6)

11. Secondary Outcome: BOTOX® Dose in Patients With Adult Focal Spasticity
Description: Adult Focal Spasticity is a condition in which muscles are continuously tight or stiff in a certain area. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 1,562 days for patients with adult focal spasticity.
Time Frame: Baseline, SV1 (up to 1,562 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 178 | 274
Units
  Baseline | 253.0 (132.6) | 346.4 (157.4)
  SV1 (N=127, 225) | 295.4 (152.4) | 355.8 (150.2)

12. Secondary Outcome: BOTOX® Dose in Patients With Cerebral Palsy
Description: Cerebral Palsy is a disability resulting in muscular incoordination and speech disturbances. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 925 days for patients with cerebral palsy.
Time Frame: Baseline, SV1 (up to 925 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 5 | 22
Units
  Baseline | 260.0 (89.4) | 245.5 (101.1)
  SV1 (N=1, 12) | 200.0 (NA) — Standard deviation is not available as only 1 patient had data at this time point. | 252.5 (105.2)

13. Secondary Outcome: BOTOX® Dose in Patients With Facial Nerve Disorder
Description: Facial nerve disorder is a condition causing twitching, weakness or paralysis of the face. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 765 days for patients with facial nerve disorder.
Time Frame: Baseline, SV1 (up to 765 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 42 | 80
Units
  Baseline | 31.3 (13.7) | 40.6 (25.4)
  SV1 (N=31, 69) | 30.9 (13.4) | 44.1 (31.2)

14. Secondary Outcome: BOTOX® Dose in Patients With "Other" Disorders
Description: "Other" disorders include focal dystonia (involuntary muscular contractions/abnormal postures), headache, pain, tics (sudden, repetitive, nonrhythmic movements/vocalizations), tremors (unintentional, rhythmic muscle movements), and other nonspecified disorders. The BOTOX® dose was assessed in this patient population. The length of time between Baseline and Subsequent Visit 1 (SV1) is scheduled at the physician's discretion and was a maximum of 568 days for patients with "other" disorders.
Time Frame: Baseline, SV1 (up to 568 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 58 | 92
Units
  Baseline | 157.2 (82.4) | 187.2 (106.8)
  SV1 (N=40, 75) | 173.4 (106.9) | 185.7 (110.1)

15. Secondary Outcome: Concurrent Procedure Resource Utilization Patterns
Description: Resource utilization patterns are assessed in terms of concurrent procedures utilized during the study (up to 1,785 days across all indications) and are grouped by highest level term. (Note: NEC=not elsewhere classified)
Time Frame: Up to 1,785 days
Population: Enrolled Cohort: All patients enrolled in the study
Measure: Number; unit: Patients
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 506 | 866
Patients
  Bone and joint therapeutic procedures | 0 | 3
  Economic and housing issues | 2 | 1
  Eye therapeutic procedures | 1 | 0
  Lifestyle issues | 3 | 9
  Therapeutic procedures and supportive care NEC | 41 | 69

16. Secondary Outcome: Concurrent Surgical Procedure Resource Utilization Patterns
Description: Resource utilization patterns are assessed in terms of concurrent surgical procedures utilized during the study (up to 1,785 days across all indications) and are grouped by highest level term. (Note: NEC=not elsewhere classified)
Time Frame: Up to 1,785 days
Population: Enrolled Cohort: All patients enrolled in the study
Measure: Number; unit: Patients
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Number analyzed (Participants) | 506 | 866
Patients
  Bone and joint therapeutic procedures | 2 | 6
  Eye therapeutic procedures | 1 | 2
  Gastrointestinal therapeutic procedures | 0 | 1
  Head and neck therapeutic procedures | 0 | 1
  Nervous system, skull&spine therapeutic procedures | 2 | 6
  Renal/urinary tract investigations & urinalyses | 1 | 0
  Renal and urinary tract therapeutic procedures | 0 | 1
  Skin appendage conditions | 0 | 1
  Soft tissue therapeutic procedures | 2 | 6
  Therapeutic procedures and supportive care NEC | 1 | 1
  Vascular therapeutic procedures | 0 | 1

ADVERSE EVENTS:
Description: The Safety Cohort included all subjects enrolled in the study who received at least one BOTOX® treatment. The Safety Cohort was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Naïve to Botox® Treatment | Non-naïve to Botox® Treatment
Serious Adverse Events (participants affected / at risk) | 5/506 | 33/866
Other Adverse Events (participants affected / at risk) | 0/506 | 0/866
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naïve to Botox® Treatment (N=506) | Non-naïve to Botox® Treatment (N=866)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 4
Multiple Sclerosis (Nervous system disorders) | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Death (General disorders) | 1 | 6
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Haemorrhoid Operation (Surgical and medical procedures) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Chest Pain (General disorders) | 0 | 1
Local Swelling (General disorders) | 0 | 1
Sudden Cardiac Death (General disorders) | 0 | 1
Gallbladder Disorder (Hepatobiliary disorders) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 0 | 1
Head Titubation (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Carpal Tunnel Decompression (Surgical and medical procedures) | 0 | 1
Knee Operation (Surgical and medical procedures) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Mental Disorder (Psychiatric disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Weight Decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 4 weeks from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.